CLINICAL TRIAL: NCT06493201
Title: Research Into Risk Factors for Hospitalization Following a Fall in Older Patients
Acronym: FDR-HPC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9242
Record Dates: First submitted 2024-04-04; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-04

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Older adults; Gait Analysis; Hospitalization; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every year, a considerable number of older people fall, with a variety of consequences. These falls can lead to hospitalization, with consequent adverse effects on these people, as well as a significant cost to society. The risk factors for falls themselves are well identified, but not those that lead to hospitalizations in older people who all fall. Some risk factors, such as age, cannot be modified. With a view to preventing hospitalizations in older patients who fall, The investigators aimed to identify functional, and therefore modifiable, risk factors for hospitalizations in patients who fall, such as gait parameters. The investigators hope that the results of this study will lead to early identification of the risk of hospitalization in these patients and thus to appropriate rehabilitation as early as possible to limit this risk.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 65 years old
* Patient having had at least one fall
* Patient able to walk without human assistance
* Hospitalized at the geriatrics center or seen in fall consultation at the Strasbourg University Hospital during the period from 05/01/2023 to 01/31/2024

Exclusion Criteria:

- Subject (and/or their legal representative if applicable) having expressed their (their) opposition to the reuse of their data

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient over 65 years old having had at least one fall and able to walk without human assistance
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03-08 (Estimated)

PRIMARY OUTCOMES:
Gait parameters assessed using the GAITrite® mat | The outcome measure is assessed at inclusion
  The recorded GAITrite® data consisted of:
  * gait speed : in (cm/s)
  * cadence: in (steps/min)
  * step time and cycle time : in (s)
  * step length and stride length : in (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie Aigue - CHU de Strasbourg - France, Strasbourg, France